CLINICAL TRIAL: NCT00003031
Title: An Open Randomised Comparative Multicentre Study of the Efficacy, Safety and Toleration of Voriconazole Versus Amphotericin-B in the Treatment of Acute Invasive Aspergillosis in Immunocompromised Patients
Brief Title: Comparison of Voriconazole and Amphotericin B in Treating Patients With Aspergillosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: EORTC-19961; EORTC-19961; PFIZER-150-307-000
Record Dates: First submitted 1999-11-01; First posted 2004-05-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Infection; Pulmonary Complications
Keywords: infection; pulmonary complications
MeSH Terms: conditions — Infections | interventions — amphotericin B, deoxycholate drug combination; Voriconazole

INTERVENTIONS:
Drug: amphotericin B deoxycholate
Drug: voriconazole

SUMMARY:
RATIONALE: Antifungal therapy with voriconazole or amphotericin B may be an effective treatment for aspergillosis. It is not yet known whether voriconazole is more effective than amphotericin B in treating patients with aspergillosis.

PURPOSE: Randomized phase III trial to compare the effectiveness of voriconazole with amphotericin B in treating patients with aspergillosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy, safety, and toleration of voriconazole versus amphotericin B (CAB) in the treatment of acute invasive aspergillosis in immunocompromised patients. II. Compare the efficacy, safety, and toleration of voriconazole versus CAB followed by other antifungal therapy in the treatment of acute invasive aspergillosis in immunocompromised patients. III. Compare survival in patients treated with voriconazole versus CAB with or without other antifungal therapy. IV. Investigate resource utilization in patients treated with voriconazole versus CAB with or without other antifungal therapy.

OUTLINE: This is an open label, randomized, multicenter study. Patients are stratified according to center, site of infection, underlying disease, and baseline neutrophil count. Patients are randomized to one of two treatment arms. Arm I: Patients receive voriconazole IV every 12 hours for 7-28 days and continue with oral voriconazole twice a day for a maximum total duration of 12 weeks of therapy. Arm II: Patients receive intravenous amphotericin B daily for at least 2 weeks; treatment continues for a maximum of 12 weeks. Patients discontinued from study drug treatment because of toxicity, intolerance or clinical failure may receive alternative (nonstudy) antifungal therapy. All patients are monitored for a total of 16 weeks.

PROJECTED ACCRUAL: A sufficient number of patients will be accrued so that 212 patients (106 per study arm) will be eligible for the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patient immunocompromised as the result of any of the following: Allogeneic bone marrow/peripheral stem cell transplant Autologous bone marrow/peripheral stem cell transplant Hematological malignancy (including lymphoma) Aplastic anemia and myelodysplastic syndromes (currently on immunosuppressive treatment) Solid organ transplantation (other than lung) Other solid organ malignancy (after cytotoxic chemotherapy) HIV/AIDS High dose prolonged corticosteroid therapy (at least 20 mg/day of prednisolone or equivalent for more than 3 weeks) or prolonged therapy with other immunosuppressive agents (e.g., azathioprine, methotrexate) Diagnosis of either definite or probable acute invasive aspergillosis Fungal infection represents a new episode of acute invasive aspergillosis Patients with the following are ineligible: Aspergilloma or allergic bronchopulmonary aspergillosis Chronic invasive aspergillosis Sarcoidosis CMV pneumonia

PATIENT CHARACTERISTICS: Age: 12 and over Life expectancy: At least 72 hours Hematopoietic: Not specified Hepatic: Bilirubin no greater than 5 times upper limit of normal (ULN) SGOT/SGPT no greater than 5 times ULN Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine no greater than 2.5 mg/dL Other: No history of hypersensitivity or intolerance to azole antifungal agents including miconazole, ketoconazole, fluconazole, or itraconazole No history of hypersensitivity or severe intolerance to conventional or lipid formulations of amphotericin B Not pregnant or nursing Fertile women must use effective contraception Negative pregnancy test No prior participation on this trial Not on artificial ventilation and unlikely to be extubated within 24 hours No condition that could affect patient safety, preclude evaluation of response, or make study completion unlikely

PRIOR CONCURRENT THERAPY: At least 8 weeks since prior systemic treatment with amphotericin B or itraconazole At least 2 weeks since prior systemic antifungal therapy for more than 96 hours at doses greater than 0.5 mg/kg/day for conventional or lipid formulations of amphotericin B or greater than 200 mg/day of itraconazole No concurrent drugs that are metabolized primarily by hepatic cytochrome P-450 enzymes or which induce or inhibit these enzymes, such as terfenadine, loratidine, astemizole, midazolam, triazolam, cisapride, rifampin, rifabutin, barbiturates, carbamazepine, coumarins, sulfonylureas, nivarapine, erythromycin, ritonavir, delaviridine, omeprazole, and phenytoin At least 2 weeks since prior rifampin, rifabutin, carbamazepine, or barbiturates for more than 3 days No concurrent investigational drugs other than cytotoxics, antiretroviral agents, or therapies for AIDS-related opportunistic infection No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) other than for treatment of granulocytopenia No concurrent white blood cell transfusions No concurrent systemic antifungal agents active against Aspergillus spp. (e.g., itraconazole, lipid formulations of amphotericin B, or flucytosine)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 1997-06; Primary Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Herbrecht, MD, Study Chair — Hopital Universitaire Hautepierre
Locations (74):
- Hartford Medical Group, Wethersfield, Connecticut, United States
- Australia (4):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (7):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- France (13):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - Hopital Edouard Herriot, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - CHR Hotel Dieu, Nantes
  - Hopital De L'Institut Pasteur, Paris
  - Hopital Robert Debre, Paris
  - Hotel Dieu de Paris, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Necker, Paris
  - Hopital Universitaire Hautepierre, Strasbourg
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (15):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Virchow Klinikum Humboldt Universitaet Berlin, Berlin
  - Universitaetskliniken Bonn, Bonn
  - Medizinische Klinik I, Dresden
  - Staedtische Kliniken Duisburg, Duisburg
  - Evangelisches Krankenhaus Essen Werden, Essen
  - University Medical Center, Freiburg im Breisgau
  - Martin Luther Universitaet, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Stefan Morsch Stiftung, Idar-Oberstein
  - Klinikum Grosshadern, Munich
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
  - Eberhard Karls Universitaet, Tübingen
  - Klinikum der Universitaet Ulm, Ulm
- Hungary (3):
  - Szent Laszlo Korhaz, Budapest
  - National Institute of Haematology and Immunology, Budapest
  - County Hospital, Kaposvár
- St. James's Hospital, Dublin, Ireland
- Hadassah University Hospital, Jerusalem, Israel
- Italy (7):
  - Ospedale San Orsola, Bologna
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale Maggiore Ca Granda, Milan
  - University and I.R.C.C.S. Policlinico San Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Ospedale Civile Pescara, Pescara
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
- Spain (7):
  - Hospital de Cruces, Barakaldo, Bilbao
  - Hospital Del Mar, Barcelona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital General Gregorio Maranon, Madrid
  - Hospital Universitasrio San Carlos, Madrid
  - University Hospital - Salamanca, Salamanca
  - Hospital Universidad Virgen Del Rocio, Seville
- Sweden (2):
  - Huddinge Hospital, Stockholm
  - Karolinska Hospital, Stockholm
- Switzerland (3):
  - University Hospital, Basel
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (7):
  - Birmingham Heartlands and Solihull NHS Trust (Teaching), Birmingham, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - King's College Hospital, London, England
  - University College Hospital, London, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Bournemouth Hospital, Bournemouth
  - North Manchester Healthcare NHS Trust, Manchester